CLINICAL TRIAL: NCT04228263
Title: Hydroxychloroquine for Improvement of Pregnancy Outcome in Unexplained Recurrent Miscarriage
Brief Title: Hydroxychloroquine and Unexplained Recurrent Miscarriage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Abdelrahman Mahmoud Mohammed, Assistant Lecturer, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HRP_2020
Record Dates: First submitted 2020-01-11; First posted 2020-01-14 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-12

CONDITIONS: Unexplained Recurrent Miscarriage
MeSH Terms: interventions — Hydroxychloroquine; Folic Acid; Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- hydroxychloroquine group (Other): hydroxychloroquine 400 mg preconceptional
  Interventions: Drug: Hydroxychloroquine; Drug: Folic Acid; Drug: Low-dose aspirin
- control group (Other): not receive hydroxychloroquine
  Interventions: Drug: Folic Acid; Drug: Low-dose aspirin

INTERVENTIONS:
Drug: Hydroxychloroquine — 400mg
  Arms: hydroxychloroquine group
Drug: Folic Acid — 5 mg
Drug: Low-dose aspirin — 75 mg

SUMMARY:
Recurrent miscarriage affects women of childbearing age worldwide. Vascular endothelial dysfunction and immunological impairment are associated with recurrent miscarriage To date, there is no effective or optimal therapeutic approach for these condition. Hydroxychloroquine has endothelial protective action via ant diabetic, lipid lowering, antioxidant effects or direct endothelial protection. Hydroxychloroquine is an antimalarial and immunomodulatory agent. In pregnancy, hydroxychloroquine is prescribed for inflammatory conditions associated with adverse perinatal outcomes such as systemic lupus erythematosus, antiphospholipid syndrome and placental inflammatory lesions such as chronic histiocytic intervillositis, hydroxychloroquine has therapeutic potential to improve placental function in pregnancies associated with heightened inflammation.

ELIGIBILITY:
Inclusion criteria

1. Women aged between 20- 40 years inclusive. 2. Body Mass Index (BMI) between 18.5 -35 Kg/m2 3. Had at least 2 previous miscarriage before 20 weeks 4. Women willing to conceive. 5. Regular Ovulatory cycles. 6. No anatomical or endocrine cause of recurrent pregnancy loss. 7. Women who have given their informed consent. 8. Negative antibody test for antiphospholipid syndrome (Lupus anticoagulant, Anticardiolipin IgM, IgG, B2glycoprotein) Exclusion criteria

1. Women who are already pregnant.
2. Known contraindication to a treatment by HCQ (retinopathy, hypersensitivity to chloroquine or HCQ, G6PD deficiency, acute intermittent porphyria, chronic liver or kidney insufficiency, extensive cutaneous psoriasis not controlled by local treatment, significant chronic digestive , hematologic disease epilepsy or psychotic disorders.) or known rare disorder of lactose metabolism .
3. Patient already using HCQ
4. Patient not get pregnant after 12 months of HCQ use.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 156 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2023-03-10 (Actual); Study Completion 2023-07-08 (Actual)

PRIMARY OUTCOMES:
Number of viable fetuses at 20 weeks gestation | 5 months

SECONDARY OUTCOMES:
Number of patients with miscarriage before 20 weeks | 5 months
Number of pregnancy complications such as ( FGR or preeclampsia, IUFD after 20 week gestation) | 9 months
Number of fetus with Major congenital anmalies | 9 months
Number of Live birth | 9 months
Number of Preterm delivery before 37 week gestation. | 8 months

CONTACTS AND LOCATIONS:
Locations (1):
- Abdel-rahman Mahmoud Mohammed, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided